CLINICAL TRIAL: NCT03875430
Title: Multicenter Prospective Observational Study to Investigate the Effectiveness of a Food Supplement Made of Hop in the Improvement of Menopausal Symptoms
Brief Title: Study to Investigate the Effectiveness of a Food Supplement Made of Hop in the Improvement of Menopausal Symptoms
Acronym: OLSEM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aristo Pharma Iberia (Industry)
Collaborators: Analysis and Research Network, S.L (Other)
Responsible Party: Sponsor
Other Study IDs: ARI-ME-18-01
Record Dates: First submitted 2019-03-11; First posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Menopause

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Perimenopausal: Patients in this group will take one capsule of a dietary supplement containing Humulus lupulus L.
  Interventions: Dietary Supplement: Humulus lupulus L
- Postmenopausal: Patients in this group will take one capsule of a dietary supplement containing Humulus lupulus L.
  Interventions: Dietary Supplement: Humulus lupulus L

INTERVENTIONS:
Dietary Supplement: Humulus lupulus L — Patients with this intervention will receive a dietary supplement to relieve the symptoms of menopause

SUMMARY:
This observational study will assess the effects of a dietary supplement based on Humulus Lupulus L. to relieve the symptoms of menopause in perimenopausal and postmenopausal women, by doing a follow up of the Cervantes scale and the Anxiety and depression Goldberg Scale in a period of 6 months. Participants will be allocated to dietary supplement being the difference between groups if they are perimenopausal or postmenopausal, and will attend to 3 visits (baseline, 3 months and 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Perimenopausal according to the Stages of Reproductive Aging Workshop (STRAW) or postmenopausal women between the ages of 40 and 60.
* Having moderate or severe hot flushes.
* Accepting and signing the Informed consent.

Exclusion Criteria:

* Women unable to answer the questionnaires.
* Women being treated with sulfonamides, methotrexate, triamterene, sulfasalazine, estrogens, phenytoin, anxiolytics, antidepressants, daily multivitamins, hormonal therapy, use of oral contraceptives in the last 3 months, herbal products to reduce vasomotor symptoms in the last months.
* Women in treatment and control for psychiatric pathology.
* Women with any comorbidity that could be the cause of a symptomatology coinciding but not bound to peri or post-menopause.
* Women diagnosed or with Clinical suspicion of breast cancer, endometrium or other hormone-dependent tumors, genital tract bleeding, actives thromboembolic disorders, active gall bladder illness or being lactose intolerant.
* Women being treated with antithyroid medications and other drugs like letrozole, raloxifene, bazedoxifene, bethanechol, desmopressin and calcitonin or other drugs that at investigators judgement could interfere in the study's result.
* Use of dietary supplements that include phytoestrogens (drinks or desserts based in soya) in the last month.
* Women with coronary diseases, strokes or chronic renal diseases, type 2 diabetes, deep vein thrombosis or pulmonary embolism.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women between 40 and 60 years old that attend ginecological consultation in Spain.
Sampling Method: Probability Sample
Enrollment: 443 (Estimated)
Dates: Start 2019-04-15 (Estimated); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life (QoL) - Measured with Score on the Cervantes Scale | Change from baseline, to 3 months and 6 months visit
  Score on the Cervantes Scale on quality of life.
  The scale is composed of 31 questions divided in 4 domains. Each question is punctuated from 0 to 5. And total scale result ranges from 0 to 155, where 0 corresponds to the maximun QoL value and 155 worst value.
Change in quality of life (QoL) - Measured with Score on the Cervantes Scale, domain: Menopause and Health. | Change from baseline, to 3 months and 6 months visit
  This domain of the Cervantes Scale is composed of 15 items, punctuated from 0 to 5. This domain ranges from 0 to 75, where 0 corresponds to abscence of physical symptoms, and 75 to the maximum level of physical problems.
Change in quality of life (QoL) - Measured with Score on the Cervantes Scale, domain: Sexuality. | Change from baseline, to 3 months and 6 months visit
  This domain of the Cervantes Scale is composed of 4 items, punctuated from 0 to 5. This domain ranges from 0 to 20, where 0 corresponds to abscence of sexual problems, and 20 to the maximum level of sexual problems.
Change in quality of life (QoL) - Measured with Score on the Cervantes Scale, domain: Psychic. | Change from baseline, to 3 months and 6 months visit
  This domain of the Cervantes Scale is composed of 9 items, punctuated from 0 to 5. This domain ranges from 0 to 45, where 0 corresponds to abscence of anxiety and depression problems, and 45 to the maximum level of anxiety and depression problems.
Change in quality of life (QoL) - Measured with Score on the Cervantes Scale, domain: Couple relationship. | Change from baseline, to 3 months and 6 months visit
  This domain of the Cervantes Scale is composed of 3 items, punctuated from 0 to 5. This domain ranges from 0 to 15, where 0 corresponds to abscence of relationship problems, and 15 to the maximum level of relationship problems.
Cervantes personality scale. | Measured at Baseline visit
  The scale is composed of 20 questions divided in 3 domains. Each question is punctuated from 0 to 5.
  First domain is introversion, it is comprised of 7 Items. This domain is punctuated from 0 to 10, where 0 represents a more extroverted personality and 10 more introverted.
  Second domain is emotional instability, it is comprised of 7 Items. This domain is punctuated from 0 to 35, where 0 represents more emotional stability and 35 more emotional instability.
  Third domain is sincerity, it is comprised of 6 Items. This domain is punctuated from 0 to 30, where 0 represents less sincere and 30 more most sincere.
Change in anxiety and depression - Measured with Score on the Anxiety and Depression Goldberg Scale | Change from baseline, to 3 months and 6 months visit
  The scale is composed of 18 items. Each item is punctuated from 0 to 5. And total scale result ranges from 0 to 90, where 0 corresponds to depression unlikely and more than 54 to severe depression.
Number of adverse events | Through the study, an average of 9 months.
  Number of adverse events (recorded in the investigator's CRF) to assess the tolerability/safety of the product
Compliance with treatment | 6 months
  Recount of product returned at the 3 months visit and at the 6 months visit of study.
Treatment satisfaction | Measured at the 6 months visit
  Treatment satisfaction is measured in three questions valued from 0 to 10, where 0 is considered worst and 10 better. The three questions are about:
  1. Patient satisfaction with the capsules.
  2. Patient satisfaction with the results of the treatment.
  3. Investigator satisfaction with the results of the treatment.